CLINICAL TRIAL: NCT03026114
Title: A ComPrehensive, ObservationaL Registry of Heart FaiLure With Mid-range and Preserved EjectiON Fraction
Acronym: APOLLON
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, BÜLENT ÖZLEK, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: MuglaSKU
Record Dates: First submitted 2017-01-10; First posted 2017-01-20 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention is planned in our study. — No intervention is planned in our study.

SUMMARY:
About 50% of all patients suffering from HF exhibit a reduced ejection fraction (EF ≤ 40%), termed HFrEF. The others may be classified into HF with midrange EF (HFmrEF, EF = 40-50%) or preserved ejection fraction (HFpEF, EF ≥ 50%).

Up to now, there are no large scale studies evaluating patients with HFmrEF and/or HFpEF in Turkey. Scarce data are available in the middle-east populations in general and Turkish patients in particular, who have different etiology, ethnic, cultural backgrounds and risk factors from those patients in the West. The aim of this study was to study Turkish patients with HFmrEF and HFpEF, and define their clinical characteristics and the signs and symptoms of heart failure, echocardiographic findings and medications at admission. With this national study, we will evaluate how recommendations of most recent European guidelines regarding pharmacological and non-pharmacological treatments are adopted in clinical practice. We will also evaluate the prevalence of the clinical profiles of patients with HFmrEF and HFpEF, according to the definitions proposed by the European Society of Cardiology, and to investigate their appropriateness in characterizing patients with different clinical presentations and needs.

Assessed outcomes included the causes of decompensation, use of medications, care quality indicators.

DETAILED DESCRIPTION:
Purpose:

To describe the demographic, clinical, and echocardiographic characteristics and management of outpatients heart failure (HF) with midrange ejection fraction (HFmrEF) and heart failure with preserved ejection fraction (HFpEF) followed by a representative setting of cardiology centres.

Background:

About 50% of all patients suffering from HF exhibit a reduced ejection fraction (EF ≤ 40%), termed HFrEF. The others may be classified into HF with midrange EF (HFmrEF, EF = 40-50%) or preserved ejection fraction (HFpEF, EF ≥ 50%). Presentation and pathophysiology of HFmrEF and HFpEF is heterogeneous and its management remains a challenge since evidence of therapeutic benefits on outcome is scarce. Up to now, there are no large scale studies evaluating patients with HFmrEF and/or HFpEF in Turkey.

Objective:

Several studies have been conducted in western countries differentiating features of epidemiology, treatment, and outcomes among patients with preserved and reduced EF. Scarce data are available in the middle-east populations in general and Turkish patients in particular, who have different etiology, ethnic, cultural backgrounds and risk factors from those patients in the West. The aim of this study was to study Turkish patients with HFmrEF and HFpEF, and define their clinical characteristics and the signs and symptoms of heart failure, echocardiographic findings and medications at admission. With this national study, we will evaluate how recommendations of most recent European guidelines regarding pharmacological and non-pharmacological treatments are adopted in clinical practice. We will also evaluate the prevalence of the clinical profiles of patients with HFmrEF and HFpEF, according to the definitions proposed by the European Society of Cardiology, and to investigate their appropriateness in characterizing patients with different clinical presentations and needs.

Methods:

We have designed a prospective, multicentre, national, observational study to characterize HFmrEF and HFpEF. Patients presented to cardiology outpatient clinics with signs and/or symptoms of HFmrEF and HFpEF will be screened. The eligibility criteria included patients older than 18 years with signs and/or symptoms of HF, admitted to public or private hospitals. Assessed outcomes included the causes of decompensation, use of medications, care quality indicators.

Data:

Clinical data, including the medical history, cardiovascular risk factors, and associate comorbidities, will be collected. The symptoms of patients will be graded according to NYHA classification. Blood samples will be collected for analysis of NT-pro-BNP and /or BNP, and complete laboratory investigations will performed as well. A 12-lead surface ECG will be recorded at 25 mm/s speed. Interpretation will be performed by a skilled investigator, and left ventricular hypertrophy (LVH) will considered according to Sokolow index.

Diastolic function parameters will be measured as follows: peak early diastolic filling (E) and late diastolic filling (A) velocities, E/A ratio, E deceleration time, early diastolic septal mitral annular velocity (e') (averaged from three cardiac cycles), and E/e' as an index of LV filling pressure. Left atrial volume index was calculated from apical four-and two-chamber views, using area - length formula. Diastolic dysfunction will be classified into four grades according to 2009 ASE guidelines.

Conclusion:

A ComPrehensive, ObservationaL Registry of Heart FaiLure With Mid-range and Preserved EjectiON Fraction (APOLLON) study aims to characterize baseline characteristics of patients with HFmrEF and HFpEF in Turkey.

ELIGIBILITY:
Inclusion Criteria:

1. Presentation to the hospital with clinical signs and symptoms of HF, according to the Framingham criteria.
2. Age≥ 18 years
3. BNP≥35 pg/ml and/or NT-proBNP≥125 pg/ml

Exclusion Criteria

1. Pregnancy
2. <18 years old
3. LVEF < %40
4. Cor pulmonale
5. Known infiltrative or hypertrophic obstructive cardiomyopathy or known pericardial constriction;
6. Primary hemodynamically significant uncorrected valvular heart disease, prosthetic valve disease
7. Myocardial infarction in past 90 days
8. Coronary artery bypass graft surgery in past 90 days
9. Percutaneous coronary intervention in past 30 days;
10. Heart transplant recipient;
11. Currently implanted left ventricular assist device;
12. Stroke in past 90 days;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented to cardiology outpatient clinics with signs and/or symptoms of HF will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
The prevalence and management strategies of heart failure with midrange ejection fraction (HFmrEF) and heart failure with preserved ejection fraction (HFpEF) patients among participating cardiology outpatient clinics. | Recruited and could be analysed at least 1065 patients after 3 months
  Outcomes included the causes of decompensation, use of medications, care quality indicators.

CONTACTS AND LOCATIONS:
Overall Officials: BÜLENT ÖZLEK, M.D., Principal Investigator — Mugla Sitki Kocman University Training and Research Hospital
Locations (1):
- Kahramanmaras Necip Fazıl City Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozlek B, Ozlek E, Tekinalp M, Kahraman S, Zencirkiran Agus H, Basaran O, Kaya BC, Rencuzogullari I, Mert KU, Cakir O, Osken A, Bekar L, Celik Y, Cil C, Dogan V, Celik O, Mert GO, Memic Sancar K, Sevinc S, Biteker M. Comparison of clinical characteristics of patients with heart failure and preserved ejection fraction with atrial fibrillation versus sinus rhythm: Insights from the APOLLON registry. Turk Kardiyol Dern Ars. 2020 Apr;48(3):234-245. doi: 10.5543/tkda.2019.77236. PMID 32281959
- [Derived] Ozlek B, Ozlek E, Agus HZ, Tekinalp M, Kahraman S, Cil C, Celik O, Basaran O, Dogan V, Kaya BC, Rencuzogullari I, Osken A, Bekar L, Cakir MO, Celik Y, Mert KU, Sancar KM, Sevinc S, Mert GO, Biteker M. Patients with HFpEF and HFmrEF have different clinical characteristics in Turkey: A multicenter observational study. Eur J Intern Med. 2019 Mar;61:88-95. doi: 10.1016/j.ejim.2018.11.001. Epub 2018 Nov 13. PMID 30446354
- [Derived] Ozlek B, Ozlek E, Celik O, Cil C, Dogan V, Tekinalp M, Zencirkiran Agus H, Kahraman S, Osken A, Rencuzogullari I, Tanik VO, Bekar L, Cakir MO, Kaya BC, Tibilli H, Celik Y, Basaran O, Mert KU, Sevinc S, Demirci E, Dondurmaci E, Biteker M. Rationale, Design, and Methodology of the APOLLON trial: A comPrehensive, ObservationaL registry of heart faiLure with midrange and preserved ejectiON fraction. Anatol J Cardiol. 2018 May;19(5):311-318. doi: 10.14744/AnatolJCardiol.2018.95595. PMID 29724973